CLINICAL TRIAL: NCT06853691
Title: The Effects of Glasses-Free 3D Training on Visual and Cognitive Function in Presbyopic Individuals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024KYPJ113
Record Dates: First submitted 2025-02-06; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Presbyopia
Keywords: Presbyopia; visual training; EEG; fNIRS
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The recruitment, grouping, training, and follow-up data collection of subjects were conducted by two different researchers, and the specific grouping information was announced after the end of the study. Any analysis conducted before the study was completed was only marked with simple symbols such as 1 and 2, and was marked by researchers who did not participate in data collection, sorting, and analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trail group (Experimental): Conduct 15 minutes of naked-eye 3D vision training. Twice a day, five days a week.
  Interventions: Other: glasses-free 3D visual training
- Control groups (No Intervention): The subjects watched ordinary 2D videos for 15 minutes each time, all under the same lighting conditions. This was done twice a day, five days a week.

INTERVENTIONS:
Other: glasses-free 3D visual training — Trail group Conduct 15 minutes of naked-eye 3D vision training. Twice a day, five days a week.
  Control groups The subjects watched ordinary 2D videos for 15 minutes each time, all under the same lighting conditions. This was done twice a day, five days a week.
  Arms: Trail group

SUMMARY:
This study aims to evaluate the effectiveness of glasses-free 3D visual training in improving visual function, visual comfort, and the application ability of visual functions in individuals with presbyopia. The research will assess changes in brain activity related to visual processing using Electroencephalogram(EEG)and Functional near-infrared spectroscopy(NIRS) before and after the training. By examining the impact of stereoscopic stimulation on the functional connectivity of brain regions, the study seeks to provide new insights into the rehabilitation of presbyopia and its underlying mechanisms. The goal is to offer a non-invasive and scientifically supported approach to improving presbyopia treatment, potentially advancing clinical practices and contributing to brain science and ophthalmology

DETAILED DESCRIPTION:
Presbyopia is a manifestation of aging, and the prevalence of presbyopia increases with age. About 1.7 to 2 billion people in the world have presbyopia. According to the criteria proposed by Hofstetter in 1950, presbyopia symptoms begin to appear in different individuals from the age of 40, and complete presbyopia occurs at the age of 60. With the occurrence of presbyopia, there will be a series of accompanying diseases, such as the decrease of contrast sensitivity, leading to visual discomfort. Moreover, near work is difficult and even affects daily life.

Conventional ophthalmic analysis and intervention are sufficient. Although invasive correction methods can achieve satisfactory visual quality, there is a certain surgical risk. It is necessary to consider not only the patient's general condition, but also the follow-up care. Some monocular correction at the cost of binocular stereoscopic vision will cause the damage of depth perception and seriously affect stereoscopic vision. Non-invasive methods also have certain limitations, such as glasses correction will increase the risk of falls due to the surrounding jumping and swimming effects, the effect of drugs is temporary, and will cause a series of adverse reactions. The glasses-free 3D vision training equipment is simple to operate, easy to implement the training process, and the content is variable, and no other equipment is needed. Due to the popularity of video terminals, the prevalence of electronic device related asthenopia is also increasing. In order to explore the improvement of accommodation function and the relief of asthenopia after glasses-free 3D training, a randomized controlled trial was designed. The effects of this training on the central nervous system were analyzed by electroencephalogram (EEG) and near-infrared spectroscopy (fNIRS).

The aim of this study is to evaluate the improvement of visual function, application ability of visual function, and visual comfort in patients with presbyopia through the intervention of glasses-free 3D visual training, and to evaluate the functional changes of brain visual-related areas in patients with presbyopia before and after the training combined with EEG and NIRS. To explore the effects of stereoscopic stimulation on the functional connectivity of brain regions and different frequency bands. To explore the scientific nature and effectiveness of glasses-free 3D visual training in the rehabilitation of presbyopia, to provide a new theoretical basis and method for the clinical treatment of presbyopia, and to provide more information and clues for exploring the complex stereo vision imaging mechanism in the fields of brain science and ophthalmology.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-60 years old, both sexes;
2. refractive error -6.0D to 5.0D, astigmatism <2.0D, anisometropia <4.0D;
3. binocular corrected visual acuity <0.2LogMAR;
4. stereoscopic threshold ≤100 ';
5. The subjects could understand the purpose of this study and sign the informed consent.

Exclusion Criteria:

1. after lens replacement; People with cataracts, which affect vision, have other eye conditions such that simultaneous vision is not possible;
2. using any medication known to affect accommodative function or wearing orthokeratology lenses in the past 1 month;
3. patients with severe systemic disease or severe mental illness;
4. Other situations where the investigator considers that the subject should not participate in the study for safety reasons or the interests of the patient.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-27 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Amplitude of accommodation | Baseline and after 6 and 12 weeks of training
  The push-up method combined with negative lens method was used. The measurements were completed by a comprehensive refractometer. It was performed according to the methods in Clinical Procedures for Ocular Examination 4th

SECONDARY OUTCOMES:
Asthenopia scale | Baseline and after 6 and 12 weeks of training
  The asthenopia scale consisted of 2 self-assessment items (" Do you have symptoms of asthenopia "and" does eye fatigue affect your study, work or life ") and 19 symptom items (" Do you feel discomfort around the eyes ")
Vergence facility | Baseline and after 6 and 12 weeks of training
  Vergence facility was tested using a lens flipper (3△BI/12△BO lens combination per eye) at 40cm with near correction
Accommodative convergence to accommodation(AC/A) | Baseline and after 6 and 12 weeks of training
  Accommodative response was measured by WAM-5500. Additional accommodative and vergence stimuli were provided by spherical lenses
The node efficiency | Baseline and after 6 and 12 weeks of training
  Electroencephalogram (EEG) was performed to track the electrical activity of the brain in real-time, and the node efficiency was calculated.
  Node efficiency is a metric that characterizes the efficiency of a single node in connecting with all other parts of the network. It reflects the centrality and importance of a node within the network.
Hemodynamic response functions | Baseline and after 6 and 12 weeks of training
  Functional near-infrared spectroscopy (fNIRS) was conducted to capture spatial information on cerebral blood flow and oxygenation conditions. Therefore, a hemodynamic response function was constructed through it.
Convergence accommodation to convergence(CA/C) | Baseline and after 6 and 12 weeks of training
  Accommodative response was measured by WAM-5500,Additional accommodative and vergence stimuli were provided by prisms
Functional connectivity network | Baseline and after 6 and 12 weeks of training
  Electroencephalogram (EEG) was performed to track the electrical activity of the brain in real-time, and the functional connectivity network was calculated.
  Functional connectivity represent changes in brain activity in time domain and frequency domain respectively through correlation and coherence.
Negative relative vergence | Baseline and after 6 and 12 weeks of training
  Negative relative vergence were measured by base in prism at 40cm with near correction
Positive relative vergence | Baseline and after 6 and 12 weeks of training
  Positive relative vergence were measured by base out prism at 40cm with near correction

OTHER OUTCOMES:
Accommodative facility | Baseline and after 6 and 12 weeks of training
  Accommodative facility was tested using a lens flipper (+0.5D/-0.5 D lens combination) at 1m with distance correction
Refraction and addition(near correction) | Baseline and after 6 and 12 weeks of training
  In a semi-dark room, the Subjective Refraction and addition(ADD) measurements were performed. Thus, the subjects' near correction prescription were obtained
Near point of convergence | Baseline and after 6 and 12 weeks of training
  Near point of convergence was measured using push-up method with near correction

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Opthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No